CLINICAL TRIAL: NCT06771206
Title: Evaluation of Accuracy of the Owlet OSS 3.0 Sensor in the Neonatal Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Owlet Baby Care, Inc. (Industry)
Collaborators: Children's of Alabama (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OWL PR0007
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Pulse Oximeter Validation
Keywords: Pulse oximetry; Neonates; Owlet; Accuracy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Owlet Arm (Experimental): All study participants meeting inclusion criteria with no stated exclusions will wear the Owlet OSS 3.0 Sensor during the study intervention. The Owlet OSS 3.0 Sensor may be placed continuously on a study subject for up to 48 hours with rotation to the opposite foot every 8 hours per device labeling to enable noninvasive data collection during the subject's standard of care blood draws. The Owlet base station will be activated in order to transmit readings but will not provide any external alarms or live displays during the monitoring period. No display of readings from the assigned Owlet device will be made available to the participant or the investigators during the time of data acquisition.
  Interventions: Device: Owlet pulse oximeter neonatal accuracy validation

INTERVENTIONS:
Device: Owlet pulse oximeter neonatal accuracy validation — This study specifically evaluates the Owlet pulse oximetry sensor, which is specifically designed and FDA cleared for for infants, and whose accuracy is specifically being validated in the neonate population.

SUMMARY:
The sponsor of this study, Owlet Baby Care, Inc., is comparing the accuracy of their pulse oximeter Sensor with the measurements of oxygen levels in newborns who are already being monitored with arterial blood samples. A minimum of 20, but up to 100 participants will be enrolled in a hospital environment and need to weigh 1500 grams or more. The purpose of the testing is to gather information on pulse oximeter readings taken by the Owlet OSS 3.0 Sensor and compare the readings to blood gas samples drawn by the medical staff. This will determine if the Owlet Sensor is accurate in newborns up to an age of 28 days after actual or expected delivery date.

The Owlet OSS 3.0 is the Sensor component within the Owlet Dream Sock, an over the counter, noninvasive pulse oximeter which is currently FDA cleared in infants 1-18 months and between 6 and 30lbs, meant to be used in the home environment. The Owlet Sock is a fabric wrap that secures the Sensor to a baby's foot. The Sensor estimates the baby's SpO2, pulse rate, and measures movement level, and transmits the wearer's readings to the paired Base Station via low energy BlueTooth energy.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single arm study to evaluate SpO2 performance of the Owlet OSS 3.0 pulse oximetry Sensor in the neonate population up to 44 weeks corrected gestational age using convenience sampling of arterial blood gas samples as a part of routine clinical monitoring.

The Owlet OSS 3.0 Sensor is the component of the Owlet Dream Sock (DEN220091) and BabySat (K222597), both Food and Drug Administration (FDA) cleared pulse oximeters for infants 1-18 months in 2023. This component performs the signal acquisition and analysis to estimate pulse rate and SpO2 readings.

The study will enroll between 20-100 neonates weighing a minimum of 1500g in the hospital setting with available arterial line access and arterial blood gas samples being performed as part of planned patient management. No additional blood gas samples will be taken beyond clinical care indications.

The primary outcome of the study is the accuracy of the Owlet OSS 3.0 Sensor SpO2 readings compared to simultaneous arterial saturation (SaO2) measurements from arterial blood gas samples as determined by a root mean square (ARMS) calculation.

Secondary outcomes will include:

* Bias in the Owlet OSS 3.0 Sensor SpO2 vs SaO2 defined as (Owlet OSS 3.0 Sensor SpO2 - SaO2).
* Precision of the Owlet OSS 3.0 Sensor SpO2 vs SaO2 defined as ABS (Owlet OSS 3.0 Sensor SpO2 - SaO2).

Accuracy will be stratified by a number of demographic elements, including by a 10 point skin tone scale and Individual Typology Angle (ITA) as determined by a spectrophotometer to demonstrate that the sensor technology under test can be accurate across diverse user populations.

The primary hypothesis is that the Owlet OSS 3.0 Sensor will measure SpO2 values within +/- 3% ARMS compared to SaO2 measurements.

Each study participant will have a total study exposure time of 48 hours. Each participant will be assigned to a unique Owlet device with a specific serial number which will be paired with the study subject identifier. The Owlet OSS 3.0 Sensor will be attached to a study subject's foot and SpO2 readings will be acquired at a set frequency and time-aligned with arterial blood gas sampling performed during the course of routine patient care. Study operators will be blinded to Owlet device readings. Time stamping of Owlet SpO2 readings will be achieved by a prescribed tapping of the device's Base Station which will mark the point at which readings simultaneous to the blood gas sample were recorded. SpO2 readings from the available noninvasive reference pulse oximeter will also be recorded during the time of blood gas sampling to document the subject's baseline SpO2 plateau.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 44 weeks corrected gestational age
* Weight equal or greater than 1500g
* Subjects with standard of care (SOC) arterial blood sampling line already in place at time of enrollment, with anticipated arterial blood gas measurements as part of their plan of care

Exclusion Criteria:

* Subjects with underdeveloped skin as assessed by a study investigator and/or reported by the clinical care team
* Subjects with abnormalities (e.g., limb deformities, open wounds, severe edema) at the planned application sites that would interfere with system measurements
* Potential subjects on extracorporeal membrane oxygenation (ECMO) or other mechanical circulatory support
* Arterial line is placed in a preductal position with the potential of pulmonary to systemic shunting
* Subjects undergoing cooling protocol/therapeutic hypothermia
* Subjects who are deemed too clinically unstable by the Principal Investigator (PI), sub-investigator and/or clinical care team to participate in the study.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pulse oximetry Accuracy - Root Mean Square | 48 hours
  Accuracy of the Owlet OSS 3.0 Sensor SpO2 readings compared to simultaneous arterial saturation (SaO2) measurements from arterial blood gas samples as determined by a root mean square (ARMS) calculation.

SECONDARY OUTCOMES:
Pulse oximetry Accuracy - Bias | 48 hours
  Bias in the Owlet OSS 3.0 Sensor SpO2 vs SaO2 defined as (Owlet OSS 3.0 Sensor SpO2 - SaO2).
Pulse oximetry Accuracy - Precision | 48 hours
  Precision of the Owlet OSS 3.0 Sensor SpO2 vs SaO2 defined as ABS (Owlet OSS 3.0 Sensor SpO2 - SaO2).

CONTACTS AND LOCATIONS:
Overall Officials: Gwenyth Fischer, M.D., Principal Investigator — University of Minnesota Medical Center; Michael A Brock, M.D., Principal Investigator — University of Alabama Birmingham - Children's of Alabama
Locations (2):
- United States (2):
  - University of Alabama Birmingham - Children's of Alabama, Birmingham, Alabama
  - University of Minnesota Medical Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okunlola OE, Lipnick MS, Batchelder PB, Bernstein M, Feiner JR, Bickler PE. Pulse Oximeter Performance, Racial Inequity, and the Work Ahead. Respir Care. 2022 Feb;67(2):252-257. doi: 10.4187/respcare.09795. Epub 2021 Nov 12. PMID 34772785
- [Background] Sjoding MW, Dickson RP, Iwashyna TJ, Gay SE, Valley TS. Racial Bias in Pulse Oximetry Measurement. N Engl J Med. 2020 Dec 17;383(25):2477-2478. doi: 10.1056/NEJMc2029240. No abstract available. PMID 33326721
- [Background] Wackernagel D, Blennow M, Hellstrom A. Accuracy of pulse oximetry in preterm and term infants is insufficient to determine arterial oxygen saturation and tension. Acta Paediatr. 2020 Nov;109(11):2251-2257. doi: 10.1111/apa.15225. Epub 2020 Mar 6. PMID 32043645